CLINICAL TRIAL: NCT05459519
Title: Effects of Dengzhanxixin Capsule on Platelet Function in Individuals at High Risk for Cardiovascular Disease (FUTURE): a Multi-center, Double-blinded, Randomized, Placebo-controlled Trial
Brief Title: Effects of Dengzhanxixin Capsule on Platelet Function in Individuals at High Risk for Cardiovascular Disease
Acronym: FUTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SFLX2022004
Record Dates: First submitted 2022-06-26; First posted 2022-07-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Diabetes; Hypertension; Hypercholesterolemia
Keywords: dengzhanxixin capsule; platelet function; primary prevention
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group A (Experimental): Dengzhanxixin Capsules plus Placebo Capsules
  Interventions: Drug: Dengzhanxixin Capsule plus Placebo Capsule
- Intervention group B (Experimental): Dengzhanxixin Capsules plus Placebo Capsules
  Interventions: Drug: Dengzhanxixin Capsule plus Placebo Capsule
- Control group (Placebo Comparator): Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dengzhanxixin Capsule plus Placebo Capsule — Dengzhanxixin Capsule, 0.54g (3 capsules) each time, twice daily; placebo, 1 capsule, twice daily
  Arms: Intervention group A
Drug: Placebo — Placebo, 4 capsules each time, twice daily
  Arms: Control group
Drug: Dengzhanxixin Capsule plus Placebo Capsule — Dengzhanxixin Capsule, 0.72g (4 capsules) each time, once daily; placebo, 4 capsules, once daily
  Arms: Intervention group B

SUMMARY:
The main objective of this clinical trial is to evaluate whether the antiplatelet efficacy of the Dengzhanxixin capsule is better than that of placebo in individuals at high-risk for atherosclerotic cardiovascular disease (ASCVD).

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of cardiovascular death, and one out of every ten people aged 35-75 in China is at high risk for ASCVD. Platelet activation is an important mechanism for the development of atherosclerosis. Antiplatelet therapy is important in preventing ASCVD.

Dengzhanxixin capsule is an over-the-counter Chinese traditional medicine; currently, it is mainly used for the adjuvant treatment of ischemic stroke and coronary heart disease. A study of 3143 patients with ischemic stroke found that the addition of Dengzhanshengmai capsules to the standard treatment could further reduce the risk of recurrent stroke and was well tolerated without increased risk of bleeding. Animal experiments also observed that Dengzhanxixin capsules had a clear antiplatelet effect. However, the antiplatelet function of Dengzhanxixin capsules in humans is still unclear. In addition, Dengzhanxixin capsules also have potential anti-inflammatory, lipid-lowering, anticoagulant, and antihypertensive effects.

The main objective of this study is to evaluate the antiplatelet efficacy and safety of Dengzhanxixin capsules in individuals at high-risk for ASCVD. The plan of the study is to recruit 165 subjects and the follow up is to be 10 weeks. This study has been approved by the Ethics Committee of Fuwai Hospital, Chinese Academy of Medical Sciences, Shenzhen.

ELIGIBILITY:
Inclusion Criteria:

The following three conditions must be met at the same time:

1. Age > 40 years, < 70 years
2. Meet any of the following conditions:

   i) Diabetes

   ii) LDL-C ≥ 4.9 mmol/L or TC ≥ 7.2 mmol/L

   iii) Hypertension; 1.8 mmol/L ≤ LDL-C < 2.6 mmol/L or 3.1 mmol/L ≤ TC < 4.1 mmol/L; 3 risk factors (including smoking, HDL-C < 1.0 mmol/L, ≥ 45 years for male or ≥ 55 years for female)

   iv) Hypertension; 2.6mmol/L ≤ LDL-C < 4.9mmol/L or 4.1mmol/L ≤ TC < 7.2mmol/L; with 2 or more risk factors (same risk factors as above)
3. Sign the informed consent

Exclusion Criteria:

Those who meet any of the following conditions are not eligible:

1. Diagnosed ASCVD, such as coronary heart disease, stroke and peripheral vascular disease
2. Past history of heart failure
3. History of symptomatic non-traumatic intracerebral hemorrhage at any time
4. History of gastrointestinal bleeding within the past 3 months or history of major surgery within 30 days
5. Need to use anticoagulation, antiplatelet or frequent use of non-steroidal anti-inflammatory drugs
6. Have used Dengzhanxixin or preparations containing Dengzhanxixin in the past 1 month
7. Have clear adverse reactions to Dengzhanxixin in the past
8. Active liver disease, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 2 times the upper limit of normal (ULN)
9. Chronic kidney disease, or estimated glomerular filtration rate (eGFR) <60ml/(min×1.73m2)
10. Pregnant or planning to become pregnant, or breastfeeding
11. Malignant tumors, or other serious diseases with an expected survival period of less than 1 year
12. Mental disorders or communication disorders, cognitive dysfunction, or other serious diseases that may affect participation in the study
13. Have participated in or are participating in other clinical trials in the past 1 month
14. Known poor adherence to study follow-up or study medication
15. Acute stage of disease: acute fever, acute pancreatitis, etc.

In addition, subjects will be excluded from the randomization clinic if they have any of the following situations:

1. Failure to complete the lead-in treatment
2. The occurrence of placebo-related adverse reactions

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in rate of platelet aggregation | "Day 0", "Week 8"
  inhibition of adenosine diphosphate (ADP)-induced platelet aggregation as measured by optical aggregometry at week 8.

SECONDARY OUTCOMES:
Changes in rate of platelet aggregation | "Day 0","Week 4","Week 8"
  1. inhibition of arachidonic acid (AA) and collagen (COLL) -induced platelet aggregation measured by optical aggregometry at week 8.
  2. inhibition of ADP, AA and COLL -induced platelet aggregation measured by optical aggregometry at week 4.
  3. At 4 weeks and 8 weeks from baseline, compare the differences of platelet P2Y12 response units (PRU) and aspirin response units (ARU)
  4. At 4 weeks and 8 weeks of treatment, compare the differences of P-selectin.
Changes in blood pressure | "Day 0","Week 4","Week 8"
  Changes in systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) at 4 and 8 weeks of treatment compared with baseline
Changes in serum lipid profile | "Day 0","Week 4","Week 8"
  changes in total cholesterol (mg/dL) , low-density lipoprotein cholesterol ester (mg/dL) , high-density lipoprotein cholesterol ester (mg/dL) , triglyceride (mg/dL) and lipoprotein(a) (mg/dL) at 4 and 8 weeks of treatment compared with baseline
Changes in coagulation profile | "Day 0","Week 4","Week 8"
  changes in prothrombin time (s), activated partial thromboplastin time (s), and thrombin time (s) at 4 and 8 weeks of treatment compared with baseline
Changes in fibrinogen | "Day 0","Week 4","Week 8"
  changes in fibrinogen (g/L) at 4 and 8 weeks of treatment compared with baseline
Changes in hs-CRP | "Day 0","Week 4","Week 8"
  changes in high-sensitivity C-reactive protein (mg/dL) at 4 and 8 weeks of treatment compared with baseline
Changes in IL-6 | "Day 0","Week 4","Week 8"
  changes in interleukin-6 (pg/mL) at 4 and 8 weeks of treatment compared with baseline
Changes in HbA1c(%) | "Day 0", "Week 8"
  Changes in HbA1c at 8 weeks of treatment compared with baseline
Number of Participants with safety endpoint | through study completion, an average of 8 weeks
  2) Liver-relate indicators:
  1. ALT ≥ 5 times ULN, or
  2. ALT ≥ 3 times ULN + bilirubin ≥ 2 times ULN (3) Kidney-related indicators:
  a. Serum creatinine increased by ≥50% from baseline, or b. Change in eGFR from baseline (4) Serious adverse events (5) Other adverse events related to the study drug (6) Drug discontinuation due to any reason

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zheng, Ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Jing Li, Ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, ShenZhen, China

IPD SHARING:
Plan to Share IPD: No